CLINICAL TRIAL: NCT05489081
Title: Promoting Implementation of Behavioral Classroom Interventions for Children With ADHD in Urban Schools: A Pilot Test, Aim 3
Brief Title: Implementation Strategy Resource Package for Behavioral Classroom Interventions: Pilot Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-019825; K23MH122577 (NIH)
Record Dates: First submitted 2022-08-02; First posted 2022-08-05 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Hyperactivity Disorder Symptoms
Keywords: Attention Deficit Hyperactivity Disorder; Positive Behavior Management; Positive Behavioral Interventions and Supports; Behavioral Classroom Management; Inattentive; Hyperactive; Impulsive
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: Participating teachers, and the students nested within their classroom, are randomized to one of two conditions: implementation strategy resource package or support as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation Resource Package Group (Experimental): Teachers in this group will receive an implementation support package and receive support in using it within their classroom management practice. Also within the intervention group (experimental), will be students nested in the classrooms of the teachers that are assigned to the intervention group.
  Interventions: Behavioral: Positive Behavior Management Toolkit
- Control Group (No Intervention): Within the control group (no intervention), teachers in this group will not receive the implementation support package nor extra support during the study period. They will continue to receive implementation support as usual. Also within the control group (no intervention) will be students nested in the classrooms of the teachers that are assigned to the control group.

INTERVENTIONS:
Behavioral: Positive Behavior Management Toolkit — The Positive Behavior Management Toolkit, or the implementation strategy resource package, is a set of resources provided to teachers in the intervention group that aims to support their use of positive behavior management practices in the classroom, particularly with students with hyperactive, inattentive, or impulsive behaviors.
  Other Names: Implementation Strategy Resource Package; Support School Success - Teacher Version (SSS-T)
  Arms: Implementation Resource Package Group

SUMMARY:
The purpose of this study is to pilot test for feasibility and initial promise an implementation strategy resource package that aims to support teachers in using behavioral classroom management interventions for children with hyperactive, inattentive, or impulsive behaviors. Participating teachers will be randomized to receive the resource package or support as usual and the research team will examine, a) teacher implementation of behavioral classroom interventions and b) mental health outcomes for enrolled children.

DETAILED DESCRIPTION:
Schools are an accessible and ecologically valid setting for children with hyperactivity, inattentive, or impulsive behaviors to receive evidence-based interventions to reduce symptoms and improve functioning. Behavioral classroom management interventions are well-established treatments for elementary-school age children with, but they can often be challenging for teachers to use. It is therefore important to develop and test implementation strategies in promoting teachers' use of behavioral classroom management interventions and in improving child outcomes. The purpose of this study is to pilot test for feasibility and initial promise an implementation strategy resource package that aims to support teachers in using behavioral classroom management interventions for children with hyperactive, inattentive, or impulsive behaviors. Participating teachers will be randomized to receive the resource package or support as usual and the research team will examine, a) teacher implementation of behavioral classroom interventions and b) mental health outcomes for enrolled children.

ELIGIBILITY:
Inclusion Criteria:

Teachers:

* A K-5 teacher at a participating school within the School District of Philadelphia
* Teach at a participating school
* Informed consent

Children:

* Is in a K-5 class of a participating teacher
* Nominated for participation by the participating teacher
* Identified by their participating teacher as displaying impairment related to inattention, hyperactivity or impulsivity
* Informed consent and assent if appropriate

Parents/Legal Guardians:

* Parent or legal guardian of child
* Identifies as familiar enough with the child to fill out measures about the child
* Has mental capacity to provide consent for the participation of child in the study and for their own participation in the study

Caregivers:

* Has been referred by the legal guardian as the primary caregiver that can more accurately complete the measures about the child
* Has mental capacity to provide consent for the participation of child in the study and for their own participation in the study

Exclusion Criteria:

Children:

* Special education classification of 'intellectual disability'
* Primary presenting concern of psychotic or autism spectrum disorders
* Presents as in acute risk of harm to self or others, such that participation in the study is clinically inappropriate because they warrant more intensive intervention

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn M Lawson, PhD, Principal Investigator — Children's Hospital of Philadelphia/University of Pennsylvania Perelman School of Medicine
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lawson GM, Owens JS, Mandell DS, Tavlin S, Rufe S, Lyon AR, Eiraldi R, Power TJ. Implementation resources to support teachers' use of behavioral classroom interventions: protocol of a randomized pilot trial. Pilot Feasibility Stud. 2023 Aug 25;9(1):151. doi: 10.1186/s40814-023-01381-4. PMID 37626422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Teachers were recruited from participating schools, and children were recruited from participating classrooms after teachers enrolled.
Pre-assignment Details: 53 participants (20 teachers, 33 children) were randomly assigned to either the intervention group or the control group following consent and baseline data collection. The number shown in each group reflect unique participants (both teachers and children). The overall number of baseline participants reflect the total number of teachers and children in each arm (i.e., 11 teachers and 17 children in the Implementation Resource Package Group and 9 teachers and 16 children in the control group).
Period: Overall Study
Arm/Group | Implementation Resource Package Group | Control Group
Started | 28 | 25
Teachers | 11 | 9
Students | 17 | 16
Completed | 28 | 22
Not Completed | 0 | 3
Not completed — student left classroom | 0 | 1
Not completed — teacher left school | 0 | 2

BASELINE CHARACTERISTICS:
Population: 53 participants (20 teachers, 33 children) were randomly assigned to either the intervention group or the control group following consent and baseline data collection. The number shown in each group reflect unique participants (both teachers and children). The overall number of baseline participants reflect the total number of teachers and children in each arm (i.e., 11 teachers and 17 children in the Implementation Resource Package Group and 9 teachers and 16 children in the control group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Implementation Resource Package Group | Control Group | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Categorical [Count of Participants; unit: Participants] — Population: This information is for the teacher participants only. Teachers reported their age by responding to a categorical question with age group brackets.
  Participants
    number analyzed (Participants) | 11 | 9 | 20
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 11 | 9 | 20
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This information is for the child participants only.
  years
    number analyzed (Participants) | 17 | 16 | 33
    (all) | 9.2 (1.6) | 9.3 (1.8) | 9.3 (1.7)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: This information is for the child participants only.
  Participants
    Male: number analyzed (Participants) | 17 | 16 | 33
    Male | 11 | 10 | 21
    Female: number analyzed (Participants) | 17 | 16 | 33
    Female | 5 | 5 | 10
    Unknown: number analyzed (Participants) | 17 | 16 | 33
    Unknown | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This information is for the teacher participants only.
  Participants
    number analyzed (Participants) | 11 | 9 | 20
    Female | 10 | 9 | 19
    Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This information is for the teacher participants only.
  Participants
    number analyzed (Participants) | 11 | 9 | 20
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 11 | 9 | 20
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This information is for the child participants only.
  Participants
    number analyzed (Participants) | 17 | 16 | 33
    Hispanic or Latino | 4 | 4 | 8
    Not Hispanic or Latino | 12 | 11 | 23
    Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This information is for the teacher participants only.
  Participants
    number analyzed (Participants) | 11 | 9 | 20
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 4 | 9
    White | 4 | 5 | 9
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This information is for the child participants only.
  Participants
    number analyzed (Participants) | 17 | 16 | 33
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 10 | 12 | 22
    White | 4 | 1 | 5
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 28 | 25 | 53
Years teaching experience [Mean (Standard Deviation); unit: years] — Population: This measure is for the teacher participants only.
  years
    number analyzed (Participants) | 11 | 9 | 20
    (all) | 14.6 (9.5) | 12.6 (9.8) | 13.7 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention Measure
Description: Teacher-reported total score on the Feasibility of Intervention Measure (FIM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Time Frame: Endpoint (i.e, at least 8 weeks from resource package receipt)
Population: The analytic sample is based on the 11 teachers randomized to the Implementation Resource Package group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 11 | 0
score on a scale | 4.52 (.47) |

2. Primary Outcome: Acceptability of Intervention Measure (AIM)
Description: Teacher-reported total score on the Acceptability of Intervention Measure (AIM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Time Frame: Endpoint (i.e, at least 8 weeks from resource package receipt)
Population: The analytic sample is the 11 teachers who were randomized to the Implementation Resource Package group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 11 | 0
score on a scale | 4.54 (.51) |

3. Primary Outcome: Intervention Appropriateness Measure (IAM)
Description: Teacher-reported total score on the Intervention Appropriateness Measure (IAM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Time Frame: Endpoint (i.e, at least 8 weeks from resource package receipt)
Population: The analytic sample is the 11 teachers who were randomized to the Implementation Resource Package group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 11 | 0
score on a scale | 4.48 (.56) |

4. Primary Outcome: Change in Observed Teacher Use of Behavioral Classroom Management Interventions
Description: A member of the study will conduct classroom observations to measure fidelity of teacher use of the behavioral classroom management interventions.
Time Frame: Baseline, midpoint (i.e., up to 7 weeks from resource package receipt), endpoint (i.e, at least 8 weeks from resource package receipt)
Population: This sample represents the number of teachers in each arm with non-missing baseline and endpoint classroom observation data.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 10 | 8
events per hour | 5.8 (11.0) | -.07 (1.9)

5. Primary Outcome: Change in Caregiver-reported Child Functional Impairment
Description: Caregiver-reported performance items on the National Institute for Children's Health Quality Vanderbilt Scale - Parent Version; These 7 items are rated on a 5-point scale (from 1 = Excellent to 5 = Problematic). The total score is the average of the 7 item scores (possible range: 1 through 5, where 1 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: Analysis was based on the sample of child participants with available parent-report data at baseline and endpoint.
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 13 | 16
change score | -.16 (.48) | .09 (.62)

6. Primary Outcome: Change in Teacher-reported Child Functional Impairment
Description: Teacher-reported performance items on the National Institute for Children's Health Quality Vanderbilt Scale - Teacher Version; These 8 items are rated on a 5-point scale (from 1 = Excellent to 5 = Problematic). The total score is the average of the 8 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: Analysis was based on the sample of child participants with available teacher-report data on this measure at baseline and endpoint.
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 16 | 14
change score | -.22 (.48) | -.29 (.61)

7. Primary Outcome: Change in Academic Productivity
Description: Teacher-reported Academic Productivity subscale score of the Academic Performance Rating Scale (APRS). The Academic Productivity subscale includes 12 items, each rated on a 5-point Likert scale from 1 to 5. Four items are reverse scored, and the total score is computed as the average of the 12 items (possible range: 1 through 5, where 5 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 16 | 14
change score | .20 (.38) | .17 (.44)

8. Primary Outcome: Change in Student-Teacher Relationship
Description: Teacher-reported total score on the Student-Teacher Relationship Scale - Short form, which consists of 15 items, rated on a 5-point scale (from 1 = Definitely does not apply to 5 = Definitely applies). Eight items are reverse score, and then the total score is computed as the average of the 15 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 16 | 14
change score | .46 (.62) | .48 (.81)

9. Primary Outcome: Feasibility of Research Procedures - Recruitment Numbers
Description: Number of teachers and students enrolled in the study
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 28 | 25
Participants
  Teachers | 11 | 9
  Students | 17 | 16

10. Primary Outcome: Feasibility of Research Procedures - Response Rate
Description: Percentage of parent- and teacher- report surveys completed across timepoints and conditions out of the number of students enrolled and randomized.
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: Analysis population is the number of students randomized in each arm.
Measure: Number; unit: percentage of surveys received
Units Other Than Participants: Surveys
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 17 | 16
Number analyzed (Surveys) | 68 | 64
percentage of surveys received | 94.1 | 90.6

11. Primary Outcome: Feasibility of Research Procedures - Retention Rate
Description: Percentage of participants who do not withdraw out of the number of enrolled and randomized teachers and students across conditions
Time Frame: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 28 | 25
percentage of participants | 100 | 88

12. Secondary Outcome: Change in Homework Performance
Description: Caregiver-reported student self-regulation factor on the Homework Performance Questionnaire - Parent Version for students in grades 1-5. The self-regulation factor consists of 9 items, each rated on a 4-point scale (0 = rarely/never, 1 = some of the time, 2 = most of the time, 3 = always/almost always). Four items are reverse scored, and then the self-regulation factor score is computed as the average of the 9 item scores (possible range: 0 through 3, where 3 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: Analysis was based on the sample of child participants with available parent-report data on this measure at baseline and endpoint.
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 12 | 13
change score | .037 (.49) | .029 (.51)

13. Secondary Outcome: Change in Caregiver-reported ADHD Symptoms
Description: Caregiver-reported inattention and hyperactivity/impulsivity symptom scores on the National Institute for Children's Health Quality Vanderbilt Scale - Parent Version, which consists of 18 items, rated on a 4-point scale (from 0 = Never to 3 = Very Often). The total score is calculated as the average of the 18 item scores (possible range: 0 through 3, where 0 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 15 | 14
change score | -.04 (.49) | .02 (.35)

14. Secondary Outcome: Change in Teacher-reported ADHD Symptoms
Description: Teacher-reported inattention and hyperactivity/impulsivity symptom scores on the National Institute for Children's Health Quality Vanderbilt Scale - Teacher Version, which consists of 18 items, rated on a 4-point scale (from 0 = Never to 3 = Very Often). The total score is calculated as the average of the 18 item scores (possible range: 0 through 3, where 0 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 16 | 15
change score | -.16 (.36) | -.15 (.60)

15. Secondary Outcome: Change in Academic Success
Description: Teacher-reported Academic Success subscale score of the Academic Performance rating Scale (APRS). The Academic Success subscale includes 7 items, each rated on a 5-point Likert scale from 1 to 5. One item is reverse scored, and the total score is computed as the average of the 7 items (possible range: 1 through 5, where 5 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 16 | 15
change score | .27 (.41) | .17 (.42)

16. Secondary Outcome: Change in Disruptive Direct Behavior Ratings
Description: Teacher-reported ratings on the disruptive behavior domain of Direct Behavior Rating Multi-Item Scales, which consist of 5 items on a 6-point scale (from 0 = "not a problem" to 6 = "serious problem"). The total score is computed as the average of the 5 items (possible range: 0 through 6, where 0 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 14 | 12
change score | -.90 (.87) | -.37 (1.63)

17. Other Pre Specified Outcome: Potential Mediators of Teacher Implementation Outcomes
Description: Teacher self-reported measures of habits regarding their use of behavior-specific praise. This consists of 12 items on a 5-point Likert scale (from 1 = "strongly disagree" to 5 = "strongly agree"). The total score is the average of the 12 item scores (possible range: 1 through 5, where 5 is the best possible outcome).
Time Frame: Baseline, endpoint (i.e, at least 8 weeks from resource package receipt)
Population: Analysis was based on sample of teacher participants with available and valid teacher-report data at baseline and endpoint.
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Implementation Resource Package Group | Control Group
Number analyzed (Participants) | 10 | 8
change score | .53 (.53) | .34 (.46)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored by the study team throughout each participating teacher and child's participation, which lasted for approximately 12-15 weeks from enrollment to endpoint data collection.
Description: This was a minimal risk behavioral intervention and as such, serious adverse events and all-cause mortality risks were not expected.
Arm/Group | Implementation Resource Package Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 0/28 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT05489081/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT05489081/ICF_000.pdf